CLINICAL TRIAL: NCT01698515
Title: Oral Health Assessment in Rheumatoid Arthritis and Other Autoimmune Diseases-- Anti- TNF Substudy
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Other Study IDs: OHARA_1898
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Anti-TNF subgroup: anti - TNF subgroup
  20 subjects with RA, who are starting TNF inhibitors based on the decision of their treating rheumatologist, will be recruited from the clinic. Patients will be starting commercially available anti-TNF agents that have already been authorized for insurance coverage. We are not requesting anti-TNFs or other drugs specifically for patients enrolled in this study from any pharmaceutical company. Patients will also continue on their background MTX and corticosteroids if they are taking these agents, and MTX will be required for patients taking Infliximab or Golimumab as per approved indication. No medications will be supplied through the study.
  --------------------------------------------------------------------------------

SUMMARY:
The objective of this study is to evaluate the effect of Tumor Necrosis Factor (TNF) inhibition on oral parameters in patients with RA and to examine changes in levels of proinflammatory cytokines in serum, gingival crevicular fluid (GCF), and saliva at an early time point (6-8 wk) and a later time point (14-16 wk) after the initiation of therapy in relation to concomitant assessment of Rheumatoid arthritis (RA) and oral clinical variables.

The purposes of the study are to:

1. Determine if oral periodontal parameters are affected by TNF inhibition;
2. Examine relationships between periodontal variables and RA variables with TNF inhibition;
3. Determine if there may be potential early response markers of clinical RA response seen using ultrasensitive analysis of oral or serum cytokines.

DETAILED DESCRIPTION:
20 subjects with RA, who are starting TNF inhibitors based on the decision of their treating rheumatologist, will be recruited only from the existing clinic population who receive ongoing clinical care at the Johns Hopkins Arthritis Center. No patients from outside the clinic will be recruited. No medications will be supplied through the study.

Study duration and numbers of visits: Patients will be followed through 14-16 weeks after the initiation of TNF inhibitor. Each patient will be seen for 4 visits: a screening visit, a baseline visit, a follow up visit between 6-8 weeks after TNF inhibitor initiation, and a final visit at weeks 14-16 after TNF inhibitor initiation. At each visit the procedures noted below will be performed. Should a patient discontinue the TNF inhibitor for any reason, a final assessment at the time of stopping will be requested.

Rheumatology Assessments: Subjects will complete standard clinical assessment questionnaires with age, race, demographic status, past medical and surgical history, co-morbid diseases, signs and symptoms of arthritis,. Multi-dimensional Health Assessment Questionnaire (MD-HAQ) and short form survey (SF)-36. Baseline joint counts for swollen, tender, and deformed or operated joints will be recorded. A Schirmer test to measure conjunctival tear production will be performed.

Oral Health and Periodontal Evaluation: Subjects will have a comprehensive oral health and periodontal evaluation. Subjects will complete standardized oral health questionnaires to assess dental health (including caries, tooth loss, periodontitis, dry mouth, and TMD) dental hygiene practices, prior dental procedures, , smoking, and access to dental care. Subjects will undergo a comprehensive dental evaluation including oral mucosal assessment, including plaque, gingivitis, and periodontal indices recorded at 6 sites per tooth, as well as an evaluation for xerostomia and temporomandibular joint (TMJ) function. Gingival crevicular fluid will be collected on paper points placed into the periodontal sulcus of the 2 most severely affected teeth and 2 sites with the least amount of periodontal inflammation. Unstimulated saliva will be collected over 5 minutes following GCF collection.

Laboratory Assessments: At each visit the investigators will obtain blood to be assayed for C-reactive protein (CRP) and other biomarkers. These will include the evaluation of a panel of inflammatory cytokines that will be tested in the blood, saliva, and GCF, to determine how these may change over time in response to TNF antagonist therapy for RA. .

Withdrawal Criteria: Patients may withdraw consent at any time and no longer participate in the oral examinations or other assessments. Patients who discontinue TNF agents for reasons of tolerability or lack of efficacy will be asked to return for a study termination visit for a follow up oral examination.

ELIGIBILITY:
INCLUSION CRITERIA:

* Adult patients age 18-75, able to provide written informed consent
* Diagnosis of RA by 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) Criteria
* Patients will not be required to be taking MTX unless they are being prescribed infliximab or golimumab as per approved indications. If taking background MTX, dose must be stable in 4 weeks and be expected to continue at the same dose for 3 months. Patients taking other nonbiological DMARDS will be excluded (leflunomide, hydroxychloroquine, sulfasalazine)
* Prednisone greater than or equal to 10 mg/day
* No prior treatment with a TNF inhibitor or other biological DMARD
* Starting anti-TNF agents with documented insurance authorization for coverage. The decision to start TNF agent and choice of particular agent will be based on the opinion of the treating rheumatologist.
* Standard starting dosing of agents will be:
* Infliximab (Remicade) 3 mg/kg IV; baseline, 2 wk, 6 wk, then q 8 wk
* Golimumab (Simponi) 50 mg subcutaneous (SC) q month
* Etanercept (Enbrel) 50 mg SC q week
* Adalimumab (Humira) 40 mg SC q every other week
* Certolizumab (Cimzia) 400 mg SC baseline, 2 wk, 4 week, then 200 mg q every other week or 400 mg q month.
* If it has been decided to use any other dosing regimen than those above, the patient will be excluded from participation.
* At least 14 teeth in the functional dentition
* Willing to practice contraception for the duration of the study period (as would be recommended to most patients starting these medications including MTX).
* Are considered eligible for a TNF inhibitor according to the following tuberculosis (TB) screening criteria:
* Have no history of latent or active TB prior to screening.
* Have no signs or symptoms suggestive of active TB upon medical history and/or physical examination.
* Have had no recent close contact with a person with active TB.
* Have a negative (greater than 5mm induration) purified protein derivative (PPD) test within 6 weeks. Patients with a positive PPD will not be allowed to enroll regardless of exposure history or receipt of Bacille Calmette-Guérin (BCG).

EXCLUSION CRITERIA:

* Taking other nonbiological DMARD unless discontinued for at least 1 month: (sulfasalazine, hydroxychloroquine, leflunomide).
* Used systemic or oral topical antibiotics (inc. tetracyclines) within 30 d of enrollment.
* Taken phenytoin, cyclosporine, or coumadin within 3 months
* Known bleeding diathesis or coagulopathy
* Subjects with valvular heart disease, joint prosthesis, or other condition requiring routine antibiotic prophylaxis for dental procedures will not necessarily be excluded unless they are not willing to receive standard appropriate antibiotic prophylaxis before dental evaluations.
* No planned elective surgery within 4 months
* Comorbid condition that in the opinion of the investigator would preclude administration of a TNF inhibitor or the performance of oral examinations
* History of latent or active granulomatous infection, including tuberculosis, histoplasmosis, or coccidiomycosis prior to screening.
* History of positive PPD or other TB exclusions noted above.
* History of persistently indeterminate on repeat exams, Quantiferon TB Gold or other gamma-interferon releasing TB assays.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 subjects with RA, who are starting TNF inhibitors based on the decision of their treating rheumatologist, will be recruited from the clinic. Patients will be starting commercially available anti-TNF agents that have already been authorized for insurance coverage. The investigators are not requesting anti-TNFs or other drugs specifically for patients enrolled in this study from Janssen or any other pharmaceutical company. Patients will also continue on their background MTX and corticosteroids if they are taking these agents, and MTX will be required for patients taking Infliximab or Golimumab as per approved indication. No medications will be supplied through the study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clifton O Bingham, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Arthritis Center, Baltimore, Maryland, United States